CLINICAL TRIAL: NCT00574288
Title: Daratumumab (HuMax®-CD38) Safety Study in Multiple Myeloma - Open Label, Dose-escalation Followed by Open Label, Single-arm Study
Brief Title: Daratumumab (HuMax®-CD38) Safety Study in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101876; GEN501 (Other: Janssen Research & Development, LLC); DARA-GEN501 (Other: Janssen Research & Development, LLC); 2007-003783-22 (EudraCT Number)
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; Safety; HuMax-CD38; Dose-escalation
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Methylprednisolone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation: Daratumumab (Experimental)
  Interventions: Drug: Part 1: Daratumumab; Other: Methylprednisolone
- Dose Expansion: Daratumumab (Experimental)
  Interventions: Drug: Part 2: Daratumumab; Other: Methylprednisolone; Other: Dexamethasone

INTERVENTIONS:
Drug: Part 1: Daratumumab — First participant will receive intravenous (injection of a substance into a vein) 0.005 milligram per kilogram (mg/kg) (planned dose) infusion of daratumumab and other participants will receive different doses. The participants will receive 7 full infusions of daratumumab and 2 predose infusions every 2 weeks. The dose of daratumumab will be escalated sequentially and considering the safety and efficacy of dose in Part 1, dose for Part 2 of the study will be decided. A predose infusion of 10% of the full dose of daratumumab will be administered a day before the first 2 full infusions.
  Other Names: HuMax-CD38
  Arms: Dose Escalation: Daratumumab
Drug: Part 2: Daratumumab — In Part 2, the participants will receive dose of daratumumab as determined in part 1 (16 mg/kg) of the study. Participants will receive 8 full infusions at weekly intervals followed by biweekly (every 2 weeks) infusions for 16 additional weeks and monthly infusions until disease progression or unmanageable toxicity, whichever comes first. Predose was dropped at some point in Part 2. A predose infusion of 10 mg daratumumab will be administered on the day before the first full infusion in select cohorts.
  Other Names: HuMax-CD38
  Arms: Dose Expansion: Daratumumab
Other: Methylprednisolone — Pre-dose: Participants (part 1) will receive methylprednisolone 80 mg intravenous (IV) injection 30 minutes to 2 hours before treatment. Participants (part 2) will receive 100 mg methylprednisolone IV 60 minutes to 2 hours before treatment; if a patient experiences no significant infusion-related reactions, the dose of methylprednisolone may be decreased to 50 mg after Visit 4.
  Post-dose: All participants (part 1) will receive 40 mg methylprednisolone orally on the first and the second day after all full infusions. During Part 2, all participants will receive 20-25 mg methylprednisolone orally or equivalent on the first and second days after all full-dose infusions.
Other: Dexamethasone — Participants (Part 2) will receive 20 mg dexamethasone intravenous (IV) injection pre-dose, on the first and second days after every full-dose infusions.
  Arms: Dose Expansion: Daratumumab

SUMMARY:
Establishment of safety profile of HuMax-CD38 when given as monotherapy in participants with multiple myeloma relapsed from or refractory to at least 2 different cytoreductive therapies and without further established treatment options.

DETAILED DESCRIPTION:
This study is conducted in two parts. In part I, participants are enrolled into cohorts at increasing dose levels. Participant safety and efficacy during part I will determine the doses used for Part II. In part II participants will be enrolled into one of two sequential treatment arms using two of the doses defined in part 1 of the study. Part II was 5 cohorts, 3 with 8 milligram per kilogram (mg/kg) and 2 with 16 mg/kg. Part I and all but the last cohort in Part II were dosed with Phase 1/ 2 drug product. The last cohort in Part II was dosed with Phase 3 drug product. Both Part I and Part II are open-label/unmasked.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of multiple myeloma (MM) requiring systemic therapy
* Age greater than or equal to (>=) 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy greater than (>) 3 months
* Relapsed from or refractory to two or more different prior therapies
* Signed Informed consent

Exclusion criteria

* Plasma cell leukemia defined as a plasma cell count > 2000/millimeter^3 (mm^3)
* Known amyloidosis
* Participants who previously have received an allogeneic stem cell transplant
* Sensory or motor neuropathy of >= grade 3
* Past or current malignancy
* Chronic or ongoing active infectious disease
* Clinically significant cardiac disease
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal (except related to MM), hepatic, hematological except MM, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
* A baseline QT interval as corrected by Fridericia's formula > 470 millisecond (msec) for female participants or > 450 msec for male participants or a complete left bundle branch block (defined as a QRS interval >= 120 msec in left bundle branch block form)
* Hypokalemia
* Clinical signs of meningeal involvement of MM
* Known severe chronic obstructive pulmonary disease or asthma defined as forced expiratory volume in 1 second (FEV1) less than (<) 60 percentage (%) of expected
* History of significant cerebrovascular disease
* Known Human Immunodeficiency Virus seropositivity
* Positive serology for hepatitis B
* Screening laboratory values
* Concomitant corticosteroid
* Other chemotherapy that is or may be active against myeloma within 3 weeks prior to Visit 2 (Part 1) or the first dose of daratumumab (Part 2). However, corticosteroid for myeloma (less than a 4-day course) could be administered within 1 week before Visit 2 (Part 1) or the first dose of daratumumab (Part 2)
* Known hypersensitivity to components of the investigational product or severe allergic or anaphylactic reactions to humanized products
* Participants who have received treatment with any nonmarket drug substance within 4 weeks before the first dose of daratumumab
* Current participation in any other interventional clinical trial
* Participants known or suspected of not being able to comply with a trial protocol (example, due to alcoholism, drug dependency, or psychological disorder)
* Breastfeeding women or women with a positive pregnancy test at Screening
* Women of childbearing potential not willing to use adequate contraception, defined as hormonal birth control or intrauterine device, during the trial and for 1 year after the last dose of daratumumab. For participants in the United States, the use of a double-barrier method is also considered adequate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-03-26 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- Boston, Massachusetts, United States
- Denmark (2):
  - Copenhagen Ø
  - Vejle
- Netherlands (2):
  - Amsterdam
  - Utrecht
- Sweden (2):
  - Huddinge
  - Lund

REFERENCES:
- [Derived] Li X, Dosne AG, Perez Ruixo C, Perez Ruixo JJ. Pharmacodynamic-Mediated Drug Disposition (PDMDD) Model of Daratumumab Monotherapy in Patients with Multiple Myeloma. Clin Pharmacokinet. 2023 May;62(5):761-777. doi: 10.1007/s40262-023-01232-8. Epub 2023 Apr 6. PMID 37022569
- [Derived] Usmani SZ, Nahi H, Plesner T, Weiss BM, Bahlis NJ, Belch A, Voorhees PM, Laubach JP, van de Donk NWCJ, Ahmadi T, Uhlar CM, Wang J, Feng H, Qi M, Richardson PG, Lonial S. Daratumumab monotherapy in patients with heavily pretreated relapsed or refractory multiple myeloma: final results from the phase 2 GEN501 and SIRIUS trials. Lancet Haematol. 2020 Jun;7(6):e447-e455. doi: 10.1016/S2352-3026(20)30081-8. PMID 32470437
- [Derived] Adams HC 3rd, Stevenaert F, Krejcik J, Van der Borght K, Smets T, Bald J, Abraham Y, Ceulemans H, Chiu C, Vanhoof G, Usmani SZ, Plesner T, Lonial S, Nijhof I, Lokhorst HM, Mutis T, van de Donk NWCJ, Sasser AK, Casneuf T. High-Parameter Mass Cytometry Evaluation of Relapsed/Refractory Multiple Myeloma Patients Treated with Daratumumab Demonstrates Immune Modulation as a Novel Mechanism of Action. Cytometry A. 2019 Mar;95(3):279-289. doi: 10.1002/cyto.a.23693. Epub 2018 Dec 11. PMID 30536810
- [Derived] Krejcik J, Frerichs KA, Nijhof IS, van Kessel B, van Velzen JF, Bloem AC, Broekmans MEC, Zweegman S, van Meerloo J, Musters RJP, Poddighe PJ, Groen RWJ, Chiu C, Plesner T, Lokhorst HM, Sasser AK, Mutis T, van de Donk NWCJ. Monocytes and Granulocytes Reduce CD38 Expression Levels on Myeloma Cells in Patients Treated with Daratumumab. Clin Cancer Res. 2017 Dec 15;23(24):7498-7511. doi: 10.1158/1078-0432.CCR-17-2027. Epub 2017 Oct 12. PMID 29025767
- [Derived] Nijhof IS, Casneuf T, van Velzen J, van Kessel B, Axel AE, Syed K, Groen RW, van Duin M, Sonneveld P, Minnema MC, Zweegman S, Chiu C, Bloem AC, Mutis T, Lokhorst HM, Sasser AK, van de Donk NW. CD38 expression and complement inhibitors affect response and resistance to daratumumab therapy in myeloma. Blood. 2016 Aug 18;128(7):959-70. doi: 10.1182/blood-2016-03-703439. Epub 2016 Jun 15. PMID 27307294
- [Derived] Lokhorst HM, Plesner T, Laubach JP, Nahi H, Gimsing P, Hansson M, Minnema MC, Lassen U, Krejcik J, Palumbo A, van de Donk NW, Ahmadi T, Khan I, Uhlar CM, Wang J, Sasser AK, Losic N, Lisby S, Basse L, Brun N, Richardson PG. Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma. N Engl J Med. 2015 Sep 24;373(13):1207-19. doi: 10.1056/NEJMoa1506348. Epub 2015 Aug 26. PMID 26308596
- See also: Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma — http://www.nejm.org/doi/full/10.1056/NEJMoa1506348

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 - <4 mg/kg: Participants were administered with 7 full intravenous (IV) infusion of 0.005, 0.05, 0.1, 0.5, 1 and 2 milligram per kilogram body weight (mg/kg) daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1 - 4 mg/kg: Participants were administered with 7 full IV infusion of 4 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1 - 8 mg/kg: Participants were administered with 7 full IV infusion of 8 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1 - 16 mg/kg: Participants were administered with 7 full IV infusion of 16 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1 - 24 mg/kg: Participants were administered with 7 full IV infusion of 24 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 2 - 8 mg/kg: Participants were administered with 8 full IV infusions of 8 mg/kg daratumumab once weekly for 8 weeks, then every 2 weeks (q2w) for 16 weeks, then every 4 weeks (q4w) until the participant experienced disease progression or unmanageable toxicity whichever came first, along with this participants also received methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions.
- Part 2 - 16 mg/kg: Participants were administered with 8 full IV infusions of 16 mg/kg daratumumab once weekly for 7 weeks, then every 2 weeks (q2w) for 14 weeks, then every 4 weeks (q4w) until the participant experienced disease progression or unmanageable toxicity whichever came first, along with this participants also received methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
Period: Overall Study
Arm/Group | Part 1 - <4 mg/kg | Part 1 - 4 mg/kg | Part 1 - 8 mg/kg | Part 1 - 16 mg/kg | Part 1 - 24 mg/kg | Part 2 - 8 mg/kg | Part 2 - 16 mg/kg
Started | 20 | 3 | 3 | 3 | 3 | 30 | 42
Completed | 0 | 0 | 0 | 1 | 1 | 4 | 14
Not Completed | 20 | 3 | 3 | 2 | 2 | 26 | 28
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 25 | 21
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Progressive Disease | 17 | 2 | 3 | 2 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - <4 mg/kg | Part 1 - 4 mg/kg | Part 1 - 8 mg/kg | Part 1 - 16 mg/kg | Part 1 - 24 mg/kg | Part 2 - 8 mg/kg | Part 2 - 16 mg/kg | Total
Number analyzed (Participants) | 20 | 3 | 3 | 3 | 3 | 30 | 42 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 2 | 2 | 3 | 2 | 21 | 22 | 63
  >=65 years | 9 | 1 | 1 | 0 | 1 | 9 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.24) | 64 (2) | 61.3 (6.11) | 53 (1.73) | 59 (9.54) | 58.6 (10.05) | 63.8 (8.27) | 61.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 0 | 0 | 0 | 9 | 15 | 33
  Male | 13 | 1 | 3 | 3 | 3 | 21 | 27 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 11 | 1 | 2 | 2 | 0 | 5 | 9 | 30
  Netherlands | 4 | 2 | 1 | 1 | 2 | 14 | 8 | 32
  Sweden | 5 | 0 | 0 | 0 | 1 | 5 | 11 | 22
  United States | 0 | 0 | 0 | 0 | 0 | 6 | 14 | 20
No. of Prior Lines of Therapy [Count of Participants; unit: Participants]
  <= 3 Lines | 2 | 2 | 0 | 0 | 0 | 6 | 16 | 26
  > 3 Lines | 18 | 1 | 3 | 3 | 3 | 24 | 26 | 78
Refractory to proteasome inhibitor (PI)/immunomodulatory agent (IMiD) [Count of Participants; unit: Participants]
  Both a PI and IMiD | 0 | 2 | 3 | 1 | 2 | 19 | 27 | 54
  PI only | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 6
  IMiD only | 0 | 0 | 0 | 1 | 1 | 6 | 4 | 12
  None | 20 | 0 | 0 | 1 | 0 | 3 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Week 28 (for Part 1) and up to approximately 2.5 years (for Part 2)
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Part 1: Daratumumab Less Than (<) 4 mg/kg: Participants were administered with 7 full intravenous (IV) infusion of 0.005, 0.05, 0.1, 0.5, 1 and 2 milligram per kilogram body weight (mg/kg) daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1: Daratumumab 4 mg/kg: Participants were administered with 7 full IV infusion of 4 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1:Daratumumab 8 mg/kg: Participants were administered with 7 full IV infusion of 8 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1: Daratumumab 16 mg/kg: Participants were administered with 8 full IV infusions of 16 mg/kg daratumumab every 2 week (q2w) for 14 weeks, then every 4 weeks (q4w), along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 1:Daratumumab 24 mg/kg: Participants were administered with 7 full IV infusion of 24 mg/kg daratumumab once weekly, along with this participants also received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
- Part 2: Daratumumab 8 mg/kg: Participants were administered with 8 full IV infusions of 8 mg/kg daratumumab once weekly for 8 weeks, then every 2 weeks (q2w) for 16 weeks, then every 4 weeks (q4w) until the participant experienced disease progression or unmanageable toxicity whichever came first, along with this participants also received methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions.
- Part 2: Daratumumab 16 mg/kg: Participants were administered with 8 full IV infusions of 16 mg/kg daratumumab once weekly for 7 weeks, then every 2 weeks (q2w) for 14 weeks, then every 4 weeks (q4w) until the participant experienced disease progression or unmanageable toxicity whichever came first, along with this participants also received methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
Arm/Group | Part 1: Daratumumab Less Than (<) 4 mg/kg | Part 1: Daratumumab 4 mg/kg | Part 1:Daratumumab 8 mg/kg | Part 1: Daratumumab 16 mg/kg | Part 1:Daratumumab 24 mg/kg | Part 2: Daratumumab 8 mg/kg | Part 2: Daratumumab 16 mg/kg
Number analyzed (Participants) | 20 | 3 | 3 | 3 | 3 | 30 | 42
participants | 19 | 3 | 3 | 3 | 3 | 30 | 41

2. Secondary Outcome: Overall Response Rate
Description: Overall response defined as percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). Per IMWG criteria, sCR: is defined as normal free light chain (FLC) ratio, and absence of clonal plasma cells (PCs) by immunohistochemistry, immunofluorescence or 2- to 4-color flow cytometry; CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5 % plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >= 90% reduction in serum M-protein plus urine M-protein level < 100mg/24 hours; PR: >= 50 % reduction of serum M-protein and reduction in 24 hour urinary M-protein by >= 90% or to <200 mg/24 hours; if the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria.
Time Frame: Up to Week 28 (for Part 1) and Week 27 (for Part 2)
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug. For Part 1, only participants treated with >= 4 mg/kg daratumumab were used for efficacy analyses and less than (<) 4 mg/kg doses were considered under the therapeutic levels.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Daratumumab 4 mg/kg | Part 1:Daratumumab 8 mg/kg | Part 1: Daratumumab 16 mg/kg | Part 1:Daratumumab 24 mg/kg | Part 2: Daratumumab 8 mg/kg | Part 2: Daratumumab 16 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 30 | 42
percentage of participants | 33.3 [0.8 to 90.6] | 0 [0 to 0] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 10.0 [2.1 to 26.5] | 35.7 [21.6 to 52.0]

3. Secondary Outcome: Part 1: Time to Response
Description: Time to first response was defined as the time from the date of first dose of daratumumab to the date of initial documentation of a response (PR or better). Time to best response was defined as the time between the date of first dose of daratumumab and the date of the initial evaluation of the best response (PR or better) to treatment. Kaplan-Meier method was used to estimate the distribution of time to response and time to best response.
Time Frame: Up to Week 28
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Daratumumab 8 mg/kg: Participants were administered with 8 mg/kg daratumumab weekly once for 8 weeks, then every 2 week (q2w) for 16 weeks, then every 4 weeks (q4w) for up to 72 weeks or until the subject experienced disease progression or unmanageable toxicity, whichever came first (possible duration of treatment: 96 weeks). Along with participants received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions.
- Daratumumab 16 mg/kg: Participants were administered with 8 full IV infusions of 16 mg/kg daratumumab once weekly for 7 weeks, then every 2 week (q2w) for 14 weeks, then every 4 weeks (q4w) for up to 72 weeks or until the subject experienced disease progression or unmanageable toxicity, whichever came first (possible duration of treatment: 96 weeks). Along with participants received methylprednisolone 80 mg IV injection before first 2 infusions and 40 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
Arm/Group | Part 1: Daratumumab 4 mg/kg | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg | Part 1:Daratumumab 24 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3
months
  Time to first response | NA [1.2 to NA] — Median and upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Median and CI was not estimable due to insufficient number of participants with events. | 8.4 [NA to NA] — Among the 3 participants on 16 mg/kg, only one participant had event, the median was set to this single uncensored value of "time to event" (defaults in PROC LIFETEST), no lower or upper bound of 95% CI calculated. | 1.9 [0.5 to 1.9]
  Time to best response | NA [1.2 to NA] — Median and upper limit of CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Median and CI was not estimable due to insufficient number of participants with events. | 8.4 [NA to NA] — Among the 3 participants on 16 mg/kg, only one participant had event, the median was set to this single uncensored value of "time to event" (defaults in PROC LIFETEST), no lower or upper bound of 95% CI calculated. | 1.9 [0.5 to 1.9]

4. Secondary Outcome: Part 2: Time to Progression (TTP)
Description: TTP was defined as the number of days from the date of first infusion (Day 1) to the date of first record of disease progression. Disease progression (IMWG criteria): increase of 25 percent (%) from lowest response level in Serum M-component and/or (the absolute increase must be >=0.5 g/dL); urine M-component and/or (the absolute increase must be >=200 mg/24 hour; only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels (absolute increase must be >10 mg/dL); Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder. Median TTP was estimated by using the Kaplan-Meier method.
Time Frame: Up to Week 27
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Daratumumab 8 mg/kg: Participants were administered with 8 mg/kg daratumumab weekly once for 8 weeks, then every 2 week (q2w) for 16 weeks, then every 4 weeks (q4w) for up to 72 weeks or until the subject experienced disease progression or unmanageable toxicity, whichever came first (possible duration of treatment: 96 weeks). Along with methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions.
- Daratumumab 16 mg/kg: Participants were administered with 8 full IV infusions of 16 mg/kg daratumumab once weekly for 7 weeks, then every 2 week (q2w) for 14 weeks, then every 4 weeks (q4w) for up to 72 weeks or until the subject experienced disease progression or unmanageable toxicity, whichever came first (possible duration of treatment: 96 weeks). Along with methylprednisolone 100 mg IV before treatment and 20-25 mg methylprednisolone orally for 2 days after all full infusions. First 2 infusions were separated by 3 week washout period.
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 30 | 42
months | 2.4 [1.4 to 3.5] | 5.6 [4.7 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Part 2: Duration of Response as Assessed Using the Method of Kaplan-Meier
Description: Duration of response was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the International Myeloma Working Group (IMWG) criteria.
Time Frame: Up to Week 27
Population: Subset of All-Treated Analysis Set included those who had overall response in Part 2.
Measure: Median (Full Range); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 3 | 15
months | 6.9 [6.2 to 10.6] | NA [5.6 to NA] — Median and upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Part 2: Progression-Free Survival
Description: Progression free survival (PFS) was defined as the time between the date of first dose of daratumumab and either disease progression or death, whichever occurs first.
Time Frame: Up to Week 27
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 30 | 42
months | 2.4 [1.4 to 3.5] | 5.6 [4.2 to 8.1]

7. Secondary Outcome: Part 2: Time to Response
Description: Time to first response was defined as the time from the date of first dose of daratumumab to the date of initial documentation of a response (PR or better). Time to best response was defined as the time between the date of first dose of daratumumab and the date of the initial evaluation of the best response (PR or better) to treatment. Time to VGPR (very good partial response) was defined as the time from the date of first dose of daratumumab to the date of initial documentation of VGPR response. The Kaplan-Meier method was used to estimate time to response.
Time Frame: Up to Week 27
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug. Here 'n' (Number of Participants Analyzed) signifies number of participants analyzed at specific time point.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 30 | 42
months
  Time to first response: number analyzed (Participants) | 3 | 15
  Time to first response | 1.36 (0.774) | 1.33 (0.955)
  Time to best response: number analyzed (Participants) | 3 | 15
  Time to best response | 1.36 (0.774) | 2.46 (2.800)
  Time to VGPR or better response: number analyzed (Participants) | 0 | 4
  Time to VGPR or better response |  | 0.49 (0.000)

8. Secondary Outcome: Part 2: Overall Survival
Description: Overall Survival (OS) was defined as the number of days from administration of the first infusion (Day 1) to date of death. Median Overall Survival was estimated by using the Kaplan-Meier method.
Time Frame: Approximately 3 years
Population: All-Treated Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab 8 mg/kg | Daratumumab 16 mg/kg
Number analyzed (Participants) | 30 | 42
months | 18.2 [7.5 to 22.6] | 34.3 [19.9 to NA] — Upper limit of CI was not estimable due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to Week 28 (for Part 1) and approximately 2.5 years
Arm/Group | Part 1 - <4 mg/kg | Part 1 - 4 mg/kg | Part 1 - 8 mg/kg | Part 1 - 16 mg/kg | Part 1 - 24 mg/kg | Part 2 - 8 mg/kg | Part 2 - 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/20 | 0/3 | 1/3 | 2/3 | 2/3 | 12/30 | 16/42
Other Adverse Events (participants affected / at risk) | 19/20 | 3/3 | 3/3 | 3/3 | 3/3 | 30/30 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - <4 mg/kg (N=20) | Part 1 - 4 mg/kg (N=3) | Part 1 - 8 mg/kg (N=3) | Part 1 - 16 mg/kg (N=3) | Part 1 - 24 mg/kg (N=3) | Part 2 - 8 mg/kg (N=30) | Part 2 - 16 mg/kg (N=42)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 2
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine Release Syndrome (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metapneumovirus Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 3
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crossmatch Incompatible (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Free Haemoglobin Present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vith Nerve Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - <4 mg/kg (N=20) | Part 1 - 4 mg/kg (N=3) | Part 1 - 8 mg/kg (N=3) | Part 1 - 16 mg/kg (N=3) | Part 1 - 24 mg/kg (N=3) | Part 2 - 8 mg/kg (N=30) | Part 2 - 16 mg/kg (N=42)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0 | 1 | 3
Haemolysis (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Monocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 0 | 2 | 3
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 9 | 6
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Lip Oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 10
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 5 | 2
Chest Discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Chest Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 5
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 5
Fatigue (General disorders) | 2 | 0 | 0 | 0 | 0 | 13 | 19
Influenza Like Illness (General disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 1
Pyrexia (General disorders) | 7 | 0 | 0 | 1 | 0 | 12 | 9
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine Release Syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 4 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 7 | 16
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 8 | 11
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Electrocardiogram QT Prolonged (Investigations) | 5 | 0 | 0 | 0 | 0 | 0 | 1
Free Haemoglobin Present (Investigations) | 4 | 0 | 0 | 0 | 0 | 0 | 0
Haptoglobin Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 4
Enzyme Abnormality (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 4 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 14
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 6 | 4
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 6
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Benign Neoplasm of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 5 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 5 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 5
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 9 | 1 | 3 | 1 | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 1 | 6 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 8 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laryngitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 5
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 12 | 10
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 4 | 2
Flushing (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypertension (Vascular disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.